CLINICAL TRIAL: NCT01082341
Title: Phase 1 and Phase 2a Clinical Trial:Immunization of Human Volunteers With P. Vivax Irradiated Sporozoites
Brief Title: Immunization of Human Volunteers With P. Vivax Irradiated Sporozoites
Acronym: SPZ-Irrad
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Malaria Vaccine and Drug Development Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Asoclinic Inmunología Ltda. (Industry)
Responsible Party: Principal Investigator, Socrates Herrera Valencia, Director, Malaria Vaccine and Drug Development Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MVDC-2008-005; SPZ IRR HUMAN (Other: MVDC); 5R01HL086488-02 (NIH)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Malaria
Keywords: GCP Good Clinical Practice; IFAT Indirect Immunofluorescence antibody test; MFA Membrane Feeding Assay; N Number (typically refers to subjects); RBC Red Blood Cells; SOP Standard Operating Procedure; TBS Thick blood smear; P. Vivax; irradiated sporozoite vaccination.
MeSH Terms: conditions — Malaria | interventions — Immunization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fy(+) (Experimental): 14 Fy(+) human volunteers in the experimental group will be immunized with 1,000-2,000 P. vivax irrad-spz bites
  Interventions: Biological: Immunization with P. vivax irradiated sporozoites
- Fy(+) control (Active Comparator): Seven Fy(+) volunteers in the control group will be exposed to non-infected mosquito bites.
  Interventions: Biological: Immunization with P. vivax irradiated sporozoites
- Fy(-) (Active Comparator): Six Fy(-) volunteers will be exposed to infective mosquito bites.
  Interventions: Biological: Immunization with P. vivax irradiated sporozoites

INTERVENTIONS:
Biological: Immunization with P. vivax irradiated sporozoites — Anopheles albimanus mosquitoes will be infected by artificial membrane feeding using blood from P. vivax infected donors. Once mosquitoes are positive will be irradiated at 15000 cGy and kept in boxes until use.
  14 Fy(+) human volunteers in the experimental group will be immunized with 1,000-2,000 P. vivax irrad-spz bites. Seven Fy(+) volunteers in the control group will be exposed to non-infected mosquito bites. Six Fy(-) volunteers will be exposed to infective mosquito bites. For the challenge both the immunized and control groups will be exposed to 3 ± 1 infective mosquito bites. Volunteers will be closely monitored post infection and will be treated with antimalarials.
  Other Names: P. vivax irradiated sporozoites vaccine

SUMMARY:
It is possible to safely protect human volunteers immunized with P. vivax irradiated sporozoites from P. vivax challenge with live sporozoites.

DETAILED DESCRIPTION:
Title: Phase 1 and Phase 2a Clinical Trial: Immunization of human volunteers with P. vivax irr-spz. (Short name: Irrad-SPZ) Population 27 healthy adult volunteers, males and non-pregnant females, between 18-45 years of age, who fulfill inclusion/exclusion criteria (described below) as determined by clinical history and serological tests. Approximately 20 parasitized blood-donor volunteers will be required to infected Anopheles mosquitoes which will be used to immunize volunteers with a total of 1000-1500 infected mosquitoes, during 8-10 months. Afterwards challenge to prove protection.

Number of Sites: 2 Study Duration: 2 years. Subject Duration : Step1: 1-2 hours to blood donors; Step 2 and 3: 2 years to immunized volunteers Objectives Primary

• To assess the safety and protective efficacy of P. vivax irradiated sporozoite vaccination.

Secondary

* To determine the immune responses and duration elicited by the P. vivax challenge in human Fy(+) volunteers previously immunized with irr-spz, as compared with non-immunized human volunteers.
* To determine the immune responses and duration elicited by irr-spz immunization scheme in human Fy(+) volunteers; comparing it with the same immunization scheme with non irr-spz in Fy(-) participants, and also with controls exposed to the same mosquito bite scheme as that of immunization but using mosquitoes without parasite infection.
* To study new antigens potentially useful to induce pre-erythrocytic protection against P. vivax malaria infection

ELIGIBILITY:
Inclusion Criteria:

* • Healthy 18 to 45 years old man or non-pregnant women.

  * To have the capacity to sign an informed consent in a free and voluntary way.
  * Have an acceptable understanding of the clinical trial through the approval of a questionnaire regarding the information given in the consent process.
  * Obligatory use of adequate contra-conceptive method from beginning of recruitment and screening time up to three months after last immunization
  * Do not have chronic or acute diseases. These conditions will be determined by clinical history, physical exam and laboratory tests.
  * To accept not traveling to malaria endemic areas during the clinical trial should
  * To have telephone at home or mobile phone that permit permanent contact for follow up
  * He (she) manifest that is willing to participated during both steps of the clinical trial.

Exclusion Criteria:

* Volunteers with less than 18 old year or more than 45 old years.
* Pregnant and suckling women will be excluded. Pregnancy will be determined both by interview, and by serum B-subunit chorionic gonadotrophin testing.
* History of moderate or severe insect, or food allergies.
* G-6PD deficiency or any Hb genetic defect (for example; sickle cell disease)
* Previous malaria infection demonstrated by think smear, PCR or specific antimalarial antibodies.
* If the subject has previously participated in a malarial vaccine trial.
* Clinical record of allergies to drug or insect bites.
* Symptoms, signs or data from laboratory test that suggests to the physician any systemic disorder like renal, hepatic, cardiovascular, pulmonary, psychiatric disorders or other illnesses that could interfere with results of clinical trial or could compromise the health of the volunteer.
* To have antibodies against hepatitis C, VIH, or hepatitis B superficial antigen and/or hepatitis B core antibodies.
* To have any abnormality in the parameters assessed by blood laboratory tests. Base-line values will be established before initiation of the clinical trial.
* Presence or history of an auto-immune disease such as; Asthma, lupus, rheumatoid arthritis, Graves's disease, Hashimoto tyroiditis, and others.
* History of surgical removal of the spleen (splenectomy).
* Volunteer with medical treatment known to alter the immune system before 3 months to recruitment, such as; cortico-steroids, chemotherapeutic agents, fludarabine, cyclosporine, tacrolimus, mycophenolate mofetil, rapamycine, ATG, alemtuzumab.
* Alcoholism or drug abuse that may interfere with social relationship of individual.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Three groups are considered to be intervened. Experimental, Control and Fy(-) groups. Comparison will be done between E and C groups for protective efficacy. For immune response tests E vs Fy(-),E vs Fy(-), and Fy(-) vs C, pairs will be compared. | 2 years

SECONDARY OUTCOMES:
The number of subjects reporting any AEs, the occurrence of specifics AEs, and discontinuation due to AEs will be tabulated. Frequency of AEs will be cross-tabulated by group for each immunization session | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Socrates Herrera, MD, Principal Investigator — Malaria Vaccine Develepment Center
Locations (1):
- Malaria Vaccine of Develepmente Center, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Wang R, Arevalo-Herrera M, Gardner MJ, Bonelo A, Carlton JM, Gomez A, Vera O, Soto L, Vergara J, Bidwell SL, Domingo A, Fraser CM, Herrera S. Immune responses to Plasmodium vivax pre-erythrocytic stage antigens in naturally exposed Duffy-negative humans: a potential model for identification of liver-stage antigens. Eur J Immunol. 2005 Jun;35(6):1859-68. doi: 10.1002/eji.200425807. PMID 15864779
- [Background] Coban C, Ishii KJ, Horii T, Akira S. Manipulation of host innate immune responses by the malaria parasite. Trends Microbiol. 2007 Jun;15(6):271-8. doi: 10.1016/j.tim.2007.04.003. Epub 2007 Apr 26. PMID 17466521
- [Background] Hoffman SL, Goh LM, Luke TC, Schneider I, Le TP, Doolan DL, Sacci J, de la Vega P, Dowler M, Paul C, Gordon DM, Stoute JA, Church LW, Sedegah M, Heppner DG, Ballou WR, Richie TL. Protection of humans against malaria by immunization with radiation-attenuated Plasmodium falciparum sporozoites. J Infect Dis. 2002 Apr 15;185(8):1155-64. doi: 10.1086/339409. Epub 2002 Apr 1. PMID 11930326
- [Background] Richie TL, Saul A. Progress and challenges for malaria vaccines. Nature. 2002 Feb 7;415(6872):694-701. doi: 10.1038/415694a. PMID 11832958
- [Background] Doolan DL, Hoffman SL, Southwood S, Wentworth PA, Sidney J, Chesnut RW, Keogh E, Appella E, Nutman TB, Lal AA, Gordon DM, Oloo A, Sette A. Degenerate cytotoxic T cell epitopes from P. falciparum restricted by multiple HLA-A and HLA-B supertype alleles. Immunity. 1997 Jul;7(1):97-112. doi: 10.1016/s1074-7613(00)80513-0. PMID 9252123
- [Background] Mellouk S, Lunel F, Sedegah M, Beaudoin RL, Druilhe P. Protection against malaria induced by irradiated sporozoites. Lancet. 1990 Mar 24;335(8691):721. doi: 10.1016/0140-6736(90)90832-p. No abstract available. PMID 1969073
- [Background] Nussenzweig R, Vanderberg J, Most H. Protective immunity produced by the injection of x-irradiated sporozoites of Plasmodium berghei. IV. Dose response, specificity and humoral immunity. Mil Med. 1969 Sep;134(10):1176-82. No abstract available. PMID 4987036
- [Background] Seguin MC, Klotz FW, Schneider I, Weir JP, Goodbary M, Slayter M, Raney JJ, Aniagolu JU, Green SJ. Induction of nitric oxide synthase protects against malaria in mice exposed to irradiated Plasmodium berghei infected mosquitoes: involvement of interferon gamma and CD8+ T cells. J Exp Med. 1994 Jul 1;180(1):353-8. doi: 10.1084/jem.180.1.353. PMID 7516412
- [Background] Weiss WR. Host-parasite interactions and immunity to irradiated sporozoites. Immunol Lett. 1990 Aug;25(1-3):39-42. doi: 10.1016/0165-2478(90)90088-8. PMID 2283161
- [Background] Weiss WR, Sedegah M, Beaudoin RL, Miller LH, Good MF. CD8+ T cells (cytotoxic/suppressors) are required for protection in mice immunized with malaria sporozoites. Proc Natl Acad Sci U S A. 1988 Jan;85(2):573-6. doi: 10.1073/pnas.85.2.573. PMID 2963334
- [Background] Collins WE, Contacos PG. Immunization of monkeys against Plasmodium cynomolgi by X-irradiated sporozoites. Nat New Biol. 1972 Apr 12;236(67):176-7. doi: 10.1038/newbio236176a0. No abstract available. PMID 4624244
- [Background] Collins WE, Nussenzweig RS, Ballou WR, Ruebush TK 2nd, Nardin EH, Chulay JD, Majarian WR, Young JF, Wasserman GF, Bathurst I, et al. Immunization of Saimiri sciureus boliviensis with recombinant vaccines based on the circumsporozoite protein of Plasmodium vivax. Am J Trop Med Hyg. 1989 May;40(5):455-64. doi: 10.4269/ajtmh.1989.40.455. PMID 2658634
- [Background] Gwadz RW, Cochrane AH, Nussenzweig V, Nussenzweig RS. Preliminary studies on vaccination of rhesus monkeys with irradiated sporozoites of Plasmodium knowlesi and characterization of surface antigens of these parasites. Bull World Health Organ. 1979;57 Suppl 1(Suppl):165-73. PMID 120766
- [Background] Zavala F, Cochrane AH, Nardin EH, Nussenzweig RS, Nussenzweig V. Circumsporozoite proteins of malaria parasites contain a single immunodominant region with two or more identical epitopes. J Exp Med. 1983 Jun 1;157(6):1947-57. doi: 10.1084/jem.157.6.1947. PMID 6189951
- [Background] Egan JE, Hoffman SL, Haynes JD, Sadoff JC, Schneider I, Grau GE, Hollingdale MR, Ballou WR, Gordon DM. Humoral immune responses in volunteers immunized with irradiated Plasmodium falciparum sporozoites. Am J Trop Med Hyg. 1993 Aug;49(2):166-73. doi: 10.4269/ajtmh.1993.49.166. PMID 8357078
- [Background] Clyde DF. Immunity to falciparum and vivax malaria induced by irradiated sporozoites: a review of the University of Maryland studies, 1971-75. Bull World Health Organ. 1990;68 Suppl(Suppl):9-12. PMID 2094597
- [Background] Clyde DF, McCarthy VC, Miller RM, Hornick RB. Specificity of protection of man immunized against sporozoite-induced falciparum malaria. Am J Med Sci. 1973 Dec;266(6):398-403. doi: 10.1097/00000441-197312000-00001. No abstract available. PMID 4590095
- [Background] Clyde DF, Most H, McCarthy VC, Vanderberg JP. Immunization of man against sporozite-induced falciparum malaria. Am J Med Sci. 1973 Sep;266(3):169-77. doi: 10.1097/00000441-197309000-00002. No abstract available. PMID 4583408
- [Background] Clyde DF. Immunization of man against falciparum and vivax malaria by use of attenuated sporozoites. Am J Trop Med Hyg. 1975 May;24(3):397-401. doi: 10.4269/ajtmh.1975.24.397. PMID 808142
- [Background] Rieckmann KH. Human immunization with attenuated sporozoites. Bull World Health Organ. 1990;68 Suppl(Suppl):13-6. PMID 2094578
- [Background] Rieckmann KH, Beaudoin RL, Cassells JS, Sell KW. Use of attenuated sporozoites in the immunization of human volunteers against falciparum malaria. Bull World Health Organ. 1979;57 Suppl 1(Suppl):261-5. PMID 120773
- [Background] Rieckmann KH, Carson PE, Beaudoin RL, Cassells JS, Sell KW. Letter: Sporozoite induced immunity in man against an Ethiopian strain of Plasmodium falciparum. Trans R Soc Trop Med Hyg. 1974;68(3):258-9. doi: 10.1016/0035-9203(74)90129-1. No abstract available. PMID 4608063
- [Background] Herrington D, Davis J, Nardin E, Beier M, Cortese J, Eddy H, Losonsky G, Hollingdale M, Sztein M, Levine M, et al. Successful immunization of humans with irradiated malaria sporozoites: humoral and cellular responses of the protected individuals. Am J Trop Med Hyg. 1991 Nov;45(5):539-47. doi: 10.4269/ajtmh.1991.45.539. PMID 1951863
- [Background] Krzych U, Lyon JA, Jareed T, Schneider I, Hollingdale MR, Gordon DM, Ballou WR. T lymphocytes from volunteers immunized with irradiated Plasmodium falciparum sporozoites recognize liver and blood stage malaria antigens. J Immunol. 1995 Oct 15;155(8):4072-7. PMID 7561118
- [Background] Glynn JR. Infecting dose and severity of malaria: a literature review of induced malaria. J Trop Med Hyg. 1994 Oct;97(5):300-16. PMID 7932927
- [Background] Glynn JR, Collins WE, Jeffery GM, Bradley DJ. Infecting dose and severity of falciparum malaria. Trans R Soc Trop Med Hyg. 1995 May-Jun;89(3):281-3. doi: 10.1016/0035-9203(95)90540-5. PMID 7660433
- [Background] Powell RD, McNamara JV. Infection with chloroquine-resistant Plasmodium falciparum in man: prepatent periods, incubation periods, and relationships between parasitemia and the onset of fever in nonimmune persons. Ann N Y Acad Sci. 1970 Oct 30;174(2):1027-41. doi: 10.1111/j.1749-6632.1970.tb45625.x. No abstract available. PMID 4993529
- [Background] Chulay JD, Schneider I, Cosgriff TM, Hoffman SL, Ballou WR, Quakyi IA, Carter R, Trosper JH, Hockmeyer WT. Malaria transmitted to humans by mosquitoes infected from cultured Plasmodium falciparum. Am J Trop Med Hyg. 1986 Jan;35(1):66-8. doi: 10.4269/ajtmh.1986.35.66. PMID 3511753
- [Background] Bejon P, Andrews L, Andersen RF, Dunachie S, Webster D, Walther M, Gilbert SC, Peto T, Hill AV. Calculation of liver-to-blood inocula, parasite growth rates, and preerythrocytic vaccine efficacy, from serial quantitative polymerase chain reaction studies of volunteers challenged with malaria sporozoites. J Infect Dis. 2005 Feb 15;191(4):619-26. doi: 10.1086/427243. Epub 2005 Jan 7. PMID 15655787
- [Background] van Dijk MR, Douradinha B, Franke-Fayard B, Heussler V, van Dooren MW, van Schaijk B, van Gemert GJ, Sauerwein RW, Mota MM, Waters AP, Janse CJ. Genetically attenuated, P36p-deficient malarial sporozoites induce protective immunity and apoptosis of infected liver cells. Proc Natl Acad Sci U S A. 2005 Aug 23;102(34):12194-9. doi: 10.1073/pnas.0500925102. Epub 2005 Aug 15. PMID 16103357
- [Background] Hurtado S, Salas ML, Romero JF, Zapata JC, Ortiz H, Arevalo-Herrera M, Herrera S. Regular production of infective sporozoites of Plasmodium falciparum and P. vivax in laboratory-bred Anopheles albimanus. Ann Trop Med Parasitol. 1997 Jan;91(1):49-60. doi: 10.1080/00034983.1997.11813111. PMID 9093429
- [Background] Zapata JC, Perlaza BL, Hurtado S, Quintero GE, Jurado D, Gonzalez I, Druilhe P, Arevalo-Herrera M, Herrera S. Reproducible infection of intact Aotus lemurinus griseimembra monkeys by Plasmodium falciparum sporozoite inoculation. J Parasitol. 2002 Aug;88(4):723-9. doi: 10.1645/0022-3395(2002)088[0723:RIOIAL]2.0.CO;2. PMID 12197121
- [Background] Herrera, S., et al., Development of a sporozoite challenge model for Plasmodium vivax in human volunteers. . (Submitte), 2009
- [Background] Herrera, S., et al., Implication of Plasmdium vivax sporozoite challenge system in vaccine development, in International Research in Infectious Diseases. 2007. p. 53.
- [Background] Herrera S, De Plata C, Gonzalez M, Perlaza BL, Bettens F, Corradin G, Arevalo-Herrera M. Antigenicity and immunogenicity of multiple antigen peptides (MAP) containing P. vivax CS epitopes in Aotus monkeys. Parasite Immunol. 1997 Apr;19(4):161-70. doi: 10.1046/j.1365-3024.1997.d01-193.x. PMID 9149283
- [Background] Herrera S, Bonelo A, Perlaza BL, Valencia AZ, Cifuentes C, Hurtado S, Quintero G, Lopez JA, Corradin G, Arevalo-Herrera M. Use of long synthetic peptides to study the antigenicity and immunogenicity of the Plasmodium vivax circumsporozoite protein. Int J Parasitol. 2004 Dec;34(13-14):1535-46. doi: 10.1016/j.ijpara.2004.10.009. PMID 15582530
- [Background] Jordan-Villegas, A., et al., Cellular and humoral responses to Plasmodium vivax irradiated sporozoites in Aotus monkeys. (In preparation), 2007
- [Background] Hollingdale MR, Krzych U. Immune responses to liver-stage parasites: implications for vaccine development. Chem Immunol. 2002;80:97-124. doi: 10.1159/000058841. No abstract available. PMID 12058653
- [Background] Yoshida N, Nussenzweig RS, Potocnjak P, Nussenzweig V, Aikawa M. Hybridoma produces protective antibodies directed against the sporozoite stage of malaria parasite. Science. 1980 Jan 4;207(4426):71-3. doi: 10.1126/science.6985745.
- [Background] Hollingdale MR, Nardin EH, Tharavanij S, Schwartz AL, Nussenzweig RS. Inhibition of entry of Plasmodium falciparum and P. vivax sporozoites into cultured cells; an in vitro assay of protective antibodies. J Immunol. 1984 Feb;132(2):909-13. PMID 6317752
- [Background] Millet P, Chizzolini C, Pieniazek NJ, Charoenvit Y, Nakamura K, Aikawa M, Jones TR, Hoffman SL, Collins WE. A monoclonal antibody directed against the sporozoite stage of Plasmodium vivax binds to liver parenchymal cells. Immunol Lett. 1992 Aug;33(3):289-94. doi: 10.1016/0165-2478(92)90075-y. PMID 1428005
- [Background] Romero P, Maryanski JL, Corradin G, Nussenzweig RS, Nussenzweig V, Zavala F. Cloned cytotoxic T cells recognize an epitope in the circumsporozoite protein and protect against malaria. Nature. 1989 Sep 28;341(6240):323-6. doi: 10.1038/341323a0. PMID 2477703
- [Background] Tsuji M, Romero P, Nussenzweig RS, Zavala F. CD4+ cytolytic T cell clone confers protection against murine malaria. J Exp Med. 1990 Nov 1;172(5):1353-7. doi: 10.1084/jem.172.5.1353. PMID 2146361
- [Background] Tsuji M, Mombaerts P, Lefrancois L, Nussenzweig RS, Zavala F, Tonegawa S. Gamma delta T cells contribute to immunity against the liver stages of malaria in alpha beta T-cell-deficient mice. Proc Natl Acad Sci U S A. 1994 Jan 4;91(1):345-9. doi: 10.1073/pnas.91.1.345. PMID 8278391
- [Background] Renggli J, Hahne M, Matile H, Betschart B, Tschopp J, Corradin G. Elimination of P. berghei liver stages is independent of Fas (CD95/Apo-I) or perforin-mediated cytotoxicity. Parasite Immunol. 1997 Mar;19(3):145-8. doi: 10.1046/j.1365-3024.1997.d01-190.x. PMID 9106820
- [Background] Calvo-Calle JM, Hammer J, Sinigaglia F, Clavijo P, Moya-Castro ZR, Nardin EH. Binding of malaria T cell epitopes to DR and DQ molecules in vitro correlates with immunogenicity in vivo: identification of a universal T cell epitope in the Plasmodium falciparum circumsporozoite protein. J Immunol. 1997 Aug 1;159(3):1362-73. PMID 9233633
- [Background] Ferreira A, Schofield L, Enea V, Schellekens H, van der Meide P, Collins WE, Nussenzweig RS, Nussenzweig V. Inhibition of development of exoerythrocytic forms of malaria parasites by gamma-interferon. Science. 1986 May 16;232(4752):881-4. doi: 10.1126/science.3085218.
- [Background] Maheshwari RK, Czarniecki CW, Dutta GP, Puri SK, Dhawan BN, Friedman RM. Recombinant human gamma interferon inhibits simian malaria. Infect Immun. 1986 Sep;53(3):628-30. doi: 10.1128/iai.53.3.628-630.1986. PMID 3091507
- [Background] Weiss WR, Berzofsky JA, Houghten RA, Sedegah M, Hollindale M, Hoffman SL. A T cell clone directed at the circumsporozoite protein which protects mice against both Plasmodium yoelii and Plasmodium berghei. J Immunol. 1992 Sep 15;149(6):2103-9. PMID 1517574
- [Background] Sedegah M, Finkelman F, Hoffman SL. Interleukin 12 induction of interferon gamma-dependent protection against malaria. Proc Natl Acad Sci U S A. 1994 Oct 25;91(22):10700-2. doi: 10.1073/pnas.91.22.10700. PMID 7938013
- [Background] Hoffman SL, Crutcher JM, Puri SK, Ansari AA, Villinger F, Franke ED, Singh PP, Finkelman F, Gately MK, Dutta GP, Sedegah M. Sterile protection of monkeys against malaria after administration of interleukin-12. Nat Med. 1997 Jan;3(1):80-3. doi: 10.1038/nm0197-80. PMID 8986746
- [Background] Fidock DA, Gras-Masse H, Lepers JP, Brahimi K, Benmohamed L, Mellouk S, Guerin-Marchand C, Londono A, Raharimalala L, Meis JF, et al. Plasmodium falciparum liver stage antigen-1 is well conserved and contains potent B and T cell determinants. J Immunol. 1994 Jul 1;153(1):190-204. PMID 7515922
- [Background] Good MF, Pombo D, Quakyi IA, Riley EM, Houghten RA, Menon A, Alling DW, Berzofsky JA, Miller LH. Human T-cell recognition of the circumsporozoite protein of Plasmodium falciparum: immunodominant T-cell domains map to the polymorphic regions of the molecule. Proc Natl Acad Sci U S A. 1988 Feb;85(4):1199-203. doi: 10.1073/pnas.85.4.1199. PMID 2448793
- [Background] Guebre-Xabier M, Schwenk R, Krzych U. Memory phenotype CD8(+) T cells persist in livers of mice protected against malaria by immunization with attenuated Plasmodium berghei sporozoites. Eur J Immunol. 1999 Dec;29(12):3978-86. doi: 10.1002/(SICI)1521-4141(199912)29:123.0.CO;2-0. PMID 10602007
- [Background] López, J.A., et al., Immunogenicity of synthetic peptides corresponding to the nonrepeat regions of the P. falciparum circumsporozoite protein. Vaccines 96. Cold Spring Harbor Laboratory 1996: p. 255-260
- [Background] Perlaza BL, Arevalo-Herrera M, Brahimi K, Quintero G, Palomino JC, Gras-Masse H, Tartar A, Druilhe P, Herrera S. Immunogenicity of four Plasmodium falciparum preerythrocytic antigens in Aotus lemurinus monkeys. Infect Immun. 1998 Jul;66(7):3423-8. doi: 10.1128/IAI.66.7.3423-3428.1998. PMID 9632616
- [Background] Perlaza BL, Zapata C, Valencia AZ, Hurtado S, Quintero G, Sauzet JP, Brahimi K, Blanc C, Arevalo-Herrera M, Druilhe P, Herrera S. Immunogenicity and protective efficacy of Plasmodium falciparum liver-stage Ag-3 in Aotus lemurinus griseimembra monkeys. Eur J Immunol. 2003 May;33(5):1321-7. doi: 10.1002/eji.200323339. PMID 12731057
- [Background] Herrera S, Herrera MA, Certa U, Corredor A, Guerrero R. Efficiency of human Plasmodium falciparum malaria vaccine candidates in Aotus lemurinus monkeys. Mem Inst Oswaldo Cruz. 1992;87 Suppl 3:423-8. doi: 10.1590/s0074-02761992000700071. PMID 1343722
- [Background] Valderrama-Aguirre A, Quintero G, Gomez A, Castellanos A, Perez Y, Mendez F, Arevalo-Herrera M, Herrera S. Antigenicity, immunogenicity, and protective efficacy of Plasmodium vivax MSP1 PV200l: a potential malaria vaccine subunit. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):16-24. doi: 10.4269/ajtmh.2005.73.16. PMID 16291762
- [Background] Arevalo-Herrera M, Castellanos A, Yazdani SS, Shakri AR, Chitnis CE, Dominik R, Herrera S. Immunogenicity and protective efficacy of recombinant vaccine based on the receptor-binding domain of the Plasmodium vivax Duffy binding protein in Aotus monkeys. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):25-31. doi: 10.4269/ajtmh.2005.73.5_suppl.0730025. PMID 16291763
- [Background] Jordan-Villegas A, Zapata JC, Perdomo AB, Quintero GE, Solarte Y, Arevalo-Herrera M, Herrera S. Aotus lemurinus griseimembra monkeys: a suitable model for Plasmodium vivax sporozoite infection. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):10-5. doi: 10.4269/ajtmh.2005.73.10. PMID 16291761
- [Background] Herrera S, Bonelo A, Perlaza BL, Fernandez OL, Victoria L, Lenis AM, Soto L, Hurtado H, Acuna LM, Velez JD, Palacios R, Chen-Mok M, Corradin G, Arevalo-Herrera M. Safety and elicitation of humoral and cellular responses in colombian malaria-naive volunteers by a Plasmodium vivax circumsporozoite protein-derived synthetic vaccine. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):3-9. doi: 10.4269/ajtmh.2005.73.3. PMID 16291760
- [Background] Fernández, O., et al. Development of a sporozoite challenge model for Plasmodium vivax in human volunteers. in Annual meeting 54th American Society of Tropical Medicine and Hygiene. December 11-15. . 2005. Washington: Am Trop J Med. Hyg.
- [Background] Arevalo-Herrera M, Herrera S. Plasmodium vivax malaria vaccine development. Mol Immunol. 2001 Dec;38(6):443-55. doi: 10.1016/s0161-5890(01)00080-3. PMID 11741694
- [Background] Castellanos A, Arevalo-Herrera M, Restrepo N, Gulloso L, Corradin G, Herrera S. Plasmodium vivax thrombospondin related adhesion protein: immunogenicity and protective efficacy in rodents and Aotus monkeys. Mem Inst Oswaldo Cruz. 2007 Jun;102(3):411-6. doi: 10.1590/s0074-02762007005000047. PMID 17568948
- [Background] Rogers WO, Gowda K, Hoffman SL. Construction and immunogenicity of DNA vaccine plasmids encoding four Plasmodium vivax candidate vaccine antigens. Vaccine. 1999 Aug 6;17(23-24):3136-44. doi: 10.1016/s0264-410x(99)00146-2. PMID 10462250
- [Background] Stowers AW, Cioce V, Shimp RL, Lawson M, Hui G, Muratova O, Kaslow DC, Robinson R, Long CA, Miller LH. Efficacy of two alternate vaccines based on Plasmodium falciparum merozoite surface protein 1 in an Aotus challenge trial. Infect Immun. 2001 Mar;69(3):1536-46. doi: 10.1128/IAI.69.3.1536-1546.2001. PMID 11179324
- [Background] Collins WE, Kaslow DC, Sullivan JS, Morris CL, Galland GG, Yang C, Saekhou AM, Xiao L, Lal AA. Testing the efficacy of a recombinant merozoite surface protein (MSP-1(19) of Plasmodium vivax in Saimiri boliviensis monkeys. Am J Trop Med Hyg. 1999 Mar;60(3):350-6. doi: 10.4269/ajtmh.1999.60.350. PMID 10466960
- [Background] Oliveira-Ferreira J, Vargas-Serrato E, Barnwell JW, Moreno A, Galinski MR. Immunogenicity of Plasmodium vivax merozoite surface protein-9 recombinant proteins expressed in E. coli. Vaccine. 2004 May 7;22(15-16):2023-30. doi: 10.1016/j.vaccine.2003.07.021. PMID 15121316
- [Background] Yazdani SS, Shakri AR, Mukherjee P, Baniwal SK, Chitnis CE. Evaluation of immune responses elicited in mice against a recombinant malaria vaccine based on Plasmodium vivax Duffy binding protein. Vaccine. 2004 Sep 9;22(27-28):3727-37. doi: 10.1016/j.vaccine.2004.03.030. PMID 15315853
- [Background] Kocken CH, Dubbeld MA, Van Der Wel A, Pronk JT, Waters AP, Langermans JA, Thomas AW. High-level expression of Plasmodium vivax apical membrane antigen 1 (AMA-1) in Pichia pastoris: strong immunogenicity in Macaca mulatta immunized with P. vivax AMA-1 and adjuvant SBAS2. Infect Immun. 1999 Jan;67(1):43-9. doi: 10.1128/IAI.67.1.43-49.1999. PMID 9864194
- [Background] Malkin EM, Durbin AP, Diemert DJ, Sattabongkot J, Wu Y, Miura K, Long CA, Lambert L, Miles AP, Wang J, Stowers A, Miller LH, Saul A. Phase 1 vaccine trial of Pvs25H: a transmission blocking vaccine for Plasmodium vivax malaria. Vaccine. 2005 May 2;23(24):3131-8. doi: 10.1016/j.vaccine.2004.12.019. PMID 15837212
- [Background] Hisaeda H, Stowers AW, Tsuboi T, Collins WE, Sattabongkot JS, Suwanabun N, Torii M, Kaslow DC. Antibodies to malaria vaccine candidates Pvs25 and Pvs28 completely block the ability of Plasmodium vivax to infect mosquitoes. Infect Immun. 2000 Dec;68(12):6618-23. doi: 10.1128/IAI.68.12.6618-6623.2000. PMID 11083773
- [Background] Arevalo-Herrera M, Solarte Y, Zamora F, Mendez F, Yasnot MF, Rocha L, Long C, Miller LH, Herrera S. Plasmodium vivax: transmission-blocking immunity in a malaria-endemic area of Colombia. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):38-43. doi: 10.4269/ajtmh.2005.73.5_suppl.0730038. PMID 16291765
- [Background] Manzano, M.R., et al., Standardization of Anopheles albimanus infection with Plasmodium vivax for sporozoite challenge of naive volunteers. (In preparation), 2009.
- [Background] Snounou G. Detection and identification of the four malaria parasite species infecting humans by PCR amplification. Methods Mol Biol. 1996;50:263-91. doi: 10.1385/0-89603-323-6:263. No abstract available. PMID 8751365
- [Background] Baird JK, Tiwari T, Martin GJ, Tamminga CL, Prout TM, Tjaden J, Bravet PP, Rawlins S, Ferrel M, Carucci D, Hoffman SL. Chloroquine for the treatment of uncomplicated malaria in Guyana. Ann Trop Med Parasitol. 2002 Jun;96(4):339-48. doi: 10.1179/000349802125001023. PMID 12171615
- [Background] Ryan JR, Stoute JA, Amon J, Dunton RF, Mtalib R, Koros J, Owour B, Luckhart S, Wirtz RA, Barnwell JW, Rosenberg R. Evidence for transmission of Plasmodium vivax among a duffy antigen negative population in Western Kenya. Am J Trop Med Hyg. 2006 Oct;75(4):575-81. PMID 17038676
- [Background] Arevalo-Herrera M, Roggero MA, Gonzalez JM, Vergara J, Corradin G, Lopez JA, Herrera S. Mapping and comparison of the B-cell epitopes recognized on the Plasmodium vivax circumsporozoite protein by immune Colombians and immunized Aotus monkeys. Ann Trop Med Parasitol. 1998 Jul;92(5):539-51. PMID 9797827
- [Background] Herrera S, Escobar P, de Plata C, Avila GI, Corradin G, Herrera MA. Human recognition of T cell epitopes on the Plasmodium vivax circumsporozoite protein. J Immunol. 1992 Jun 15;148(12):3986-90. PMID 1376347
- [Background] Arevalo-Herrera M, Valencia AZ, Vergara J, Bonelo A, Fleischhauer K, Gonzalez JM, Restrepo JC, Lopez JA, Valmori D, Corradin G, Herrera S. Identification of HLA-A2 restricted CD8(+) T-lymphocyte responses to Plasmodium vivax circumsporozoite protein in individuals naturally exposed to malaria. Parasite Immunol. 2002 Mar;24(3):161-9. doi: 10.1046/j.1365-3024.2002.00449.x. PMID 12078650
- [Background] Perlaza BL, Sauzet JP, Balde AT, Brahimi K, Tall A, Corradin G, Druilhe P. Long synthetic peptides encompassing the Plasmodium falciparum LSA3 are the target of human B and T cells and are potent inducers of B helper, T helper and cytolytic T cell responses in mice. Eur J Immunol. 2001 Jul;31(7):2200-9. doi: 10.1002/1521-4141(200107)31:73.0.co;2-l. PMID 11449374
- [Background] Miller LH, Mason SJ, Dvorak JA, McGinniss MH, Rothman IK. Erythrocyte receptors for (Plasmodium knowlesi) malaria: Duffy blood group determinants. Science. 1975 Aug 15;189(4202):561-3. doi: 10.1126/science.1145213.
- [Background] Herrera S, Gomez A, Vera O, Vergara J, Valderrama-Aguirre A, Maestre A, Mendez F, Wang R, Chitnis CE, Yazdani SS, Arevalo-Herrera M. Antibody response to Plasmodium vivax antigens in Fy-negative individuals from the Colombian Pacific coast. Am J Trop Med Hyg. 2005 Nov;73(5 Suppl):44-9. doi: 10.4269/ajtmh.2005.73.44. PMID 16291766
- [Background] Ocana-Morgner C, Mota MM, Rodriguez A. Malaria blood stage suppression of liver stage immunity by dendritic cells. J Exp Med. 2003 Jan 20;197(2):143-51. doi: 10.1084/jem.20021072. PMID 12538654
- [Background] Coban C, Ishii KJ, Kawai T, Hemmi H, Sato S, Uematsu S, Yamamoto M, Takeuchi O, Itagaki S, Kumar N, Horii T, Akira S. Toll-like receptor 9 mediates innate immune activation by the malaria pigment hemozoin. J Exp Med. 2005 Jan 3;201(1):19-25. doi: 10.1084/jem.20041836. PMID 15630134
- [Background] Engwerda CR, Good MF. Interactions between malaria parasites and the host immune system. Curr Opin Immunol. 2005 Aug;17(4):381-7. doi: 10.1016/j.coi.2005.05.010. PMID 15950450
- [Background] Scheller LF, Azad AF. Maintenance of protective immunity against malaria by persistent hepatic parasites derived from irradiated sporozoites. Proc Natl Acad Sci U S A. 1995 Apr 25;92(9):4066-8. doi: 10.1073/pnas.92.9.4066. PMID 7732032
- [Background] Mueller AK, Labaied M, Kappe SH, Matuschewski K. Genetically modified Plasmodium parasites as a protective experimental malaria vaccine. Nature. 2005 Jan 13;433(7022):164-7. doi: 10.1038/nature03188. Epub 2004 Dec 5. PMID 15580261
- [Background] Mangold KA, Manson RU, Koay ES, Stephens L, Regner M, Thomson RB Jr, Peterson LR, Kaul KL. Real-time PCR for detection and identification of Plasmodium spp. J Clin Microbiol. 2005 May;43(5):2435-40. doi: 10.1128/JCM.43.5.2435-2440.2005. PMID 15872277
- [Background] Baird JK, Lacy MD, Basri H, Barcus MJ, Maguire JD, Bangs MJ, Gramzinski R, Sismadi P, Krisin, Ling J, Wiady I, Kusumaningsih M, Jones TR, Fryauff DJ, Hoffman SL; United States Naval Medical Research Unit 2 Clinical Trials Team. Randomized, parallel placebo-controlled trial of primaquine for malaria prophylaxis in Papua, Indonesia. Clin Infect Dis. 2001 Dec 15;33(12):1990-7. doi: 10.1086/324085. Epub 2001 Nov 12. PMID 11712091
- [Background] Chatterjee S, Francois G, Druilhe P, Timperman G, Wery M. Immunity to Plasmodium berghei exoerythrocytic forms derived from irradiated sporozoites. Parasitol Res. 1996;82(4):297-303. doi: 10.1007/s004360050117. PMID 8740544
- [Background] Malkin E, Dubovsky F, Moree M. Progress towards the development of malaria vaccines. Trends Parasitol. 2006 Jul;22(7):292-5. doi: 10.1016/j.pt.2006.05.002. Epub 2006 May 16. PMID 16707275
- [Background] Beier JC, Davis JR, Vaughan JA, Noden BH, Beier MS. Quantitation of Plasmodium falciparum sporozoites transmitted in vitro by experimentally infected Anopheles gambiae and Anopheles stephensi. Am J Trop Med Hyg. 1991 May;44(5):564-70. doi: 10.4269/ajtmh.1991.44.564. PMID 2063960
- [Background] Doolan DL, Hoffman SL. Pre-erythrocytic-stage immune effector mechanisms in Plasmodium spp. infections. Philos Trans R Soc Lond B Biol Sci. 1997 Sep 29;352(1359):1361-7. doi: 10.1098/rstb.1997.0121. PMID 9355128
- [Background] Doolan DL, Martinez-Alier N. Immune response to pre-erythrocytic stages of malaria parasites. Curr Mol Med. 2006 Mar;6(2):169-85. doi: 10.2174/156652406776055249. PMID 16515509
- [Background] Hoffman, S.L., et al., Attacking the infected hepatocyte. In Malaria Vaccine Development: A Multi- Immune Response Approach, ed. S.L. Hoffman. 1996, Washington, DC: ASM Press. 35-75.
- [Background] Nussenzweig RS, Vanderberg JP, Most H, Orton C. Specificity of protective immunity produced by x-irradiated Plasmodium berghei sporozoites. Nature. 1969 May 3;222(5192):488-9. doi: 10.1038/222488a0. No abstract available. PMID 5768632
- [Background] Nardin EH, Nussenzweig RS, Altszuler R, Herrington D, Levine M, Murphy J, Davis J, Bathurst I, Barr P, Romero P, et al. Cellular and humoral immune responses to a recombinant P. falciparum CS protein in sporozoite-immunized rodents and human volunteers. Bull World Health Organ. 1990;68 Suppl(Suppl):85-7. PMID 2094595
- [Background] Procell PM, Collins WE, Campbell GH. Circumsporozoite protein of the human malaria parasite Plasmodium ovale identified with monoclonal antibodies. Infect Immun. 1988 Feb;56(2):376-9. doi: 10.1128/iai.56.2.376-379.1988. PMID 3338845
- [Background] Rathore D, Nagarkatti R, Jani D, Chattopadhyay R, de la Vega P, Kumar S, McCutchan TF. An immunologically cryptic epitope of Plasmodium falciparum circumsporozoite protein facilitates liver cell recognition and induces protective antibodies that block liver cell invasion. J Biol Chem. 2005 May 27;280(21):20524-9. doi: 10.1074/jbc.M414254200. Epub 2005 Mar 21. PMID 15781464
- [Background] Cox RJ, Brokstad KA, Zuckerman MA, Wood JM, Haaheim LR, Oxford JS. An early humoral immune response in peripheral blood following parenteral inactivated influenza vaccination. Vaccine. 1994 Aug;12(11):993-9. doi: 10.1016/0264-410x(94)90334-4. PMID 7975853
- [Background] Crotty S, Aubert RD, Glidewell J, Ahmed R. Tracking human antigen-specific memory B cells: a sensitive and generalized ELISPOT system. J Immunol Methods. 2004 Mar;286(1-2):111-22. doi: 10.1016/j.jim.2003.12.015. PMID 15087226
- [Background] Malaspina A, Moir S, Orsega SM, Vasquez J, Miller NJ, Donoghue ET, Kottilil S, Gezmu M, Follmann D, Vodeiko GM, Levandowski RA, Mican JM, Fauci AS. Compromised B cell responses to influenza vaccination in HIV-infected individuals. J Infect Dis. 2005 May 1;191(9):1442-50. doi: 10.1086/429298. Epub 2005 Mar 24. PMID 15809902
- [Background] Palmer DR, Krzych U. Cellular and molecular requirements for the recall of IL-4-producing memory CD4(+)CD45RO(+)CD27(-) T cells during protection induced by attenuated Plasmodium falciparum sporozoites. Eur J Immunol. 2002 Mar;32(3):652-61. doi: 10.1002/1521-4141(200203)32:33.0.CO;2-9. PMID 11857339
- [Background] Mills KH. Regulatory T cells: friend or foe in immunity to infection? Nat Rev Immunol. 2004 Nov;4(11):841-55. doi: 10.1038/nri1485. PMID 15516964
- [Background] Di Fabio S, Mbawuike IN, Kiyono H, Fujihashi K, Couch RB, McGhee JR. Quantitation of human influenza virus-specific cytotoxic T lymphocytes: correlation of cytotoxicity and increased numbers of IFN-gamma producing CD8+ T cells. Int Immunol. 1994 Jan;6(1):11-9. doi: 10.1093/intimm/6.1.11. PMID 8148319
- [Background] Wang R, Epstein J, Baraceros FM, Gorak EJ, Charoenvit Y, Carucci DJ, Hedstrom RC, Rahardjo N, Gay T, Hobart P, Stout R, Jones TR, Richie TL, Parker SE, Doolan DL, Norman J, Hoffman SL. Induction of CD4(+) T cell-dependent CD8(+) type 1 responses in humans by a malaria DNA vaccine. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10817-22. doi: 10.1073/pnas.181123498. Epub 2001 Aug 28. PMID 11526203
- [Background] Wang R, Epstein J, Charoenvit Y, Baraceros FM, Rahardjo N, Gay T, Banania JG, Chattopadhyay R, de la Vega P, Richie TL, Tornieporth N, Doolan DL, Kester KE, Heppner DG, Norman J, Carucci DJ, Cohen JD, Hoffman SL. Induction in humans of CD8+ and CD4+ T cell and antibody responses by sequential immunization with malaria DNA and recombinant protein. J Immunol. 2004 May 1;172(9):5561-9. doi: 10.4049/jimmunol.172.9.5561. PMID 15100299
- [Background] Nijman HW, Houbiers JG, Vierboom MP, van der Burg SH, Drijfhout JW, D'Amaro J, Kenemans P, Melief CJ, Kast WM. Identification of peptide sequences that potentially trigger HLA-A2.1-restricted cytotoxic T lymphocytes. Eur J Immunol. 1993 Jun;23(6):1215-9. doi: 10.1002/eji.1830230603. PMID 7684681
- [Background] Calvo-Calle JM, Oliveira GA, Nardin EH. Human CD4+ T cells induced by synthetic peptide malaria vaccine are comparable to cells elicited by attenuated Plasmodium falciparum sporozoites. J Immunol. 2005 Dec 1;175(11):7575-85. doi: 10.4049/jimmunol.175.11.7575. PMID 16301667
- [Background] Pritchard JK, Stephens M, Donnelly P. Inference of population structure using multilocus genotype data. Genetics. 2000 Jun;155(2):945-59. doi: 10.1093/genetics/155.2.945. PMID 10835412
- [Derived] Lopez-Perez M, Jain A, Davies DH, Vasquez-Jimenez JM, Herrera SM, Onate J, Felgner PL, Herrera S, Arevalo-Herrera M. Profiling the antibody response of humans protected by immunization with Plasmodium vivax radiation-attenuated sporozoites. Sci Rep. 2024 Feb 2;14(1):2790. doi: 10.1038/s41598-024-53175-0. PMID 38307966
- [Derived] Arevalo-Herrera M, Vasquez-Jimenez JM, Lopez-Perez M, Vallejo AF, Amado-Garavito AB, Cespedes N, Castellanos A, Molina K, Trejos J, Onate J, Epstein JE, Richie TL, Herrera S. Protective Efficacy of Plasmodium vivax Radiation-Attenuated Sporozoites in Colombian Volunteers: A Randomized Controlled Trial. PLoS Negl Trop Dis. 2016 Oct 19;10(10):e0005070. doi: 10.1371/journal.pntd.0005070. eCollection 2016 Oct. PMID 27760143
- See also: www.inmuno.org — http://inmuno.org